CLINICAL TRIAL: NCT01448551
Title: Novel Individually Tailored Mobile Messages to Enhance Weight Loss for Teens
Brief Title: MPOWERed Messages: Tailored Mobile Messages to Enhance Weight Loss for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan J Woolford, MD, MPH, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F022685-1; 5K23HD058797-02 (NIH)
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Obesity; Treatment; Adolescents; Text Messages; Mobile phones; Multidisciplinary
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Messaging (Experimental)
  Interventions: Behavioral: Tailored Mobile Messages to Enhance Weight Loss for Teens
- Control (No Intervention): Participation in the MPOWER program without receiving tailored text messages

INTERVENTIONS:
Behavioral: Tailored Mobile Messages to Enhance Weight Loss for Teens — For this trial adolescents will be allowed to use their own phone (with reimbursement for any study-related costs), or will be provided with a mobile phone, if requested. Participants will receive messages delivered daily over the course of 20 weeks. The content of the messages will be tailored on participants' responses to the MPOWER enrollment survey and the initial tailoring questionnaire. On school days, all messages will be sent after 3 pm (which is after school hours for most Michigan middle and high schools). Therefore, patients will not need to carry cell phones to school. The tailored messages will utilize various degrees of personalization, adaptation and feedback - including momentary assessments with feedback requiring a text reply from the adolescents.
  Other Names: MPOWERed Messages
  Arms: Text Messaging

SUMMARY:
Obesity affects millions of American children and increases their risk of adult obesity, a myriad of serious illnesses, increased healthcare costs, and premature death. It is vital to find ways to reverse this epidemic. Multidisciplinary behavioral weight management programs offer the promise of effectively treating childhood obesity. However, participants in such programs often find it challenging to follow recommended treatment plans and frequently drop out from programs without completing them. The proposed project aims to address these problems through frequent contact with patients between office visits. This interim contact will be achieved by automatically sending tailored messages to the mobile phones of adolescents enrolled in a multidisciplinary weight management program (the MPOWER program), as an adjunct to clinic visits.

The investigators hypothesize that program participants who receive the tailored text messages will experience lower attrition rates, increased treatment adherence, and greater weight loss compared to those program participants who do not receive the messages.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 95th percentile for sex and age according to CDC growth charts
* Enrollment in the MPOWER program
* At least one parent willing and able to participate in the MPOWER program with the adolescent
* Absence of any major medical illness, disability, or moderate/severe mental disorder (e.g., liver disease, renal failure, cancer, bipolar disorder)

Exclusion Criteria:

* Presence of any major medical illness, disability, or moderate/severe mental disorder (e.g., renal failure, cancer, bipolar disorder)
* Physical, mental, or cognitive handicaps that prevent participation
* Chronic use of medications that may affect study outcomes (e.g., Diuretics, oral steroids)
* Girls who are pregnant, planning to become pregnant in the next 6 months, lactating, or within 6 months postpartum

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Session attendance | Over the course of 6 months
Adherence to MPOWER program homework assignments | Over the course of 6 months
Satisfaction with the MPOWER program | At the completion of 3 months and 6 months in the program
Drop out | Prior to completion of the 6 month program

SECONDARY OUTCOMES:
Change in body mass index | After 3 months and 6 months in the MPOWER program
Objective measurement of daily participation in moderate to vigorous activity | After 3 months and 6 months in the MPOWER program
Self-efficacy for achieving MPOWER recommendations for the 6 target behaviors | After 3 months and 6 months in the MPOWER program6 month
  Using a self-efficacy scale developed by Resnicow we will measure self-efficacy for consuming breakfast daily, achieving recommended amounts of fruits and vegetables, obtaining 60 to 90 minutes of moderate to vigorous physical activity on most days, limiting fast food consumption to no more than once per week, consuming no more than three 8 oz servings of sugar-sweetened beverages per week, and engaging in no more than 2 hours of screen time per day.
Intrinsic motivation to increase intake of fruits and vegetables and to increase physical activity | After 3 months and 6 months in the MPOWER program
  Intrinsic motivation will be measured using the Treatment Self-Regulation Questionnaire for Nutrition and the Treatment Self-Regulation Questionnaire for Physical Activity
Change in self-report of the six behaviors targeted in the intervention | After 3 months and 6 months in the MPOWER program
  The behaviors addressed are: Breakfast (self-report, in response to the question, During the last 7days, how many days did you eat breakfast?) Fruits and vegetables (24 hour food recall) Fast food (self-report in response to the question, During the last 7 days, how often did you eat food purchased at a fast food restaurant?) Sugar-sweetened beverages (24 hour food recall) Screen time (self-report in response to questions regarding number of hours of screen time per day on school days and non-school days) Physical activity (self-report using the Fitnessgram Activity log)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Woolford, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States